CLINICAL TRIAL: NCT02842359
Title: Efficacy Evaluation of Metabolic, Anti-inflammatory, and Antioxidative Factors of Irbesartan/Atorvastatin Fixed-dose Combination in Type 2 Diabetic Patients Diagnosed With Hyperlipidemia and Hypertension, With Adequately Controlled Blood Glucose Levels
Brief Title: Evaluation of the Fixed-dose Combination of Irbesartan/Atorvastatin in Type 2 Diabetic Patients Diagnosed With Hyperlipidemia and Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATOIRL07827; U1111-1182-8092 (Other: UTN)
Record Dates: First submitted 2016-07-20; First posted 2016-07-22 (Estimated); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Irbesartan; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Rovelito (Experimental): Fixed-dose combination of irbesartan/atorvastatin will be given orally daily for 28 days
  Interventions: Drug: Irbesartan/atorvastatin fixed dose combination
- Irbesartan (Active Comparator): Irbesartan will be given orally daily for 28 days
  Interventions: Drug: Irbesartan SR47436
- Atorvastatin (Active Comparator): Atorvastatin will be given orally daily for 28 days
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Irbesartan/atorvastatin fixed dose combination — Pharmaceutical form:Tablet Route of administration: Oral
  Other Names: Rovelito
  Arms: Rovelito
Drug: Irbesartan SR47436 — Pharmaceutical form:Tablet Route of administration: Oral
  Other Names: Aprovel
  Arms: Irbesartan
Drug: Atorvastatin — Pharmaceutical form:Tablet Route of administration: Oral
  Other Names: Newvast
  Arms: Atorvastatin

SUMMARY:
Primary Objective:

To evaluate the effect of irbesartan/atorvastatin fixed-dose combination comparing to each irbesartan and atorvastatin on flow mediated dilation change in type 2 diabetic patients diagnosed with hyperlipidemia, hypertension.

Secondary Objective:

To evaluate efficacy of blood pressure and hyperlipidemic factors of irbesartan/atorvastatin fixed-dose combination in type 2 diabetic patients diagnosed with hyperlipidemia and hypertension, with adequately controlled blood glucose levels in groups.

DETAILED DESCRIPTION:
The total study duration per patient is up to maximum of 7 weeks.

ELIGIBILITY:
Inclusion criteria:

* Patients aged ≥19 years to <75 years.
* Patients without medication history of hyperlipidemia and hypertension within 3 months following registration, among type 2 diabetic patients diagnosed with hyperlipidemia and stage I hypertension (systolic blood pressure: ≥140mmHg, ≤159 mmHg or diastolic blood pressure: ≥90 mmHg, ≤99mmHg), with adequately controlled hemoglobin levels.
* Patients who signed a written consent to data utilization.
* Diagnosis of diabetes:
* HemoglobinA1c ≥6.5% or;
* Fasting plasma glucose level above 8 hour ≥126 mg/dL or;
* Plasma glucose ≥200 mg/dL ( 11.1 mmol/l) 2 hours after a 75g glucose load or;
* Symptoms (such as polyuria, polydipsia, unexplained weight loss) and a random plasma glucose ≥200 mg/dL (11.1 mmol/L).

Exclusion criteria:

* Patients indicated as contraindication in the approved labeling of Rovelito.
* Pregnant/nursing women.
* Patients with difference in blood pressure systolic blood pressure ≥20 mmHg or diastolic blood pressure ≥10mmHg in the arm selected during screening at Visit 1.
* Patients who were administered Angiotensin II receptor blockers, angiotensin converting enzyme inhibitors, or HMG-CoA reductase inhibitors in 2 months.
* Patients who had taken antidiabetics in the past.
* Patients who have to or may take any drug suggested in the prohibited concomitant medications during the study period.
* Patients with tolerance or hypersensitivity to angiotensin II receptor blocker or HMGCoA reductase inhibitor, or an ingredient of this drug, or with history of multi-drug allergy.
* Patients with genetic angioedema, or medical history of angioedema when treating with angiotensin converting enzyme inhibitor or angiotensin II receptor antagonist
* Patients who have suffered from fibromyalgia, myopathy, rhabdomyolysis, or sudden arthralgia, or adverse events while taking statins in the past.
* Creatine phosphokinase (CPK) >5 times of the upper limit of normal (ULN).
* Patients diagnosed with secondary hypertension or suspected of secondary hypertension by the Investigator (coarctation of aorta, primary aldosteronism, renal artery stenosis, renal hypertension, pheochromocytoma, Cushing syndrome, etc.).
* Patients with poorly controlled hypothyroidism despite treatment
* Type 1 diabetic patients or poorly controlled type 2 diabetic patients (HemoglobinA1c ≥7.5%)
* Patients with arrhythmia requiring separate treatment.
* Patients with the following past history:
* Severe cerebrovascular disease (cerebral infarction, cerebral hemorrhage, etc.), hypertensive encephalopathy, transient ischemic attack (TIA), which occurred in the recent 6 months.
* Severe heart disease (NYHA class III-IV heart failure), clinically significant valvular disease of the heart, myocardial infarction and unstable angina in the recent 6 months.
* Angioplasty or coronary artery bypass graft (CABG) surgery.
* If patients have clinically significant renal or hepatic diseases , or significant hematologic test findings at screening (serum creatinine ≥ 2mg/dL, AST or ALT [aspartate transaminase or alanine transaminase] ≥3 times of the ULN).
* Patients suspected of pancreatitis or active gall bladder disease by the Investigator.
* Surgical or internal disease likely to significantly change absorption, distribution, metabolism, and elimination of drug, which falls under one of the followings (but not limited to):
* Major gastrointestinal surgical history such as gastrectomy, gastro-enterostomy or bowel resection, gastric bypass, gastrointestinal stapling, or gastrointestinal banding, medical history of active inflammatory bowel syndrome at present or in the past 12 months, current active gastritis, ulcer, gastrointestinal/rectal hemorrhage, or urinary tract obstruction that is deemed clinically significant by the Investigator.
* Patients with volume depletion, as clinically judged by the Investigator, using vital signs, skin turgor pressure, mucous membrane wettability, and laboratory values.
* All chronic inflammatory patients requiring chronic inflammatory treatment.
* Patients with past history of autoimmune disease, such as chronic rheumatoid arthritis, systemic lupus erythematosus, etc.
* Patients with past clinical history of alcohol or drug abuse.
* Patients with history of malignant tumors including leukemia and lymphoma in the past 5 years.
* Patients who have been administered another investigational product within 30 days prior to participation in this clinical study (from the time when they signed the informed consent form).
* Patients who may not be measured for flow mediated dilatation in Investigator's judgment for a congenital or secondary reason in the bilateral brachial artery.
* Patients who are deemed ineligible as subject in Investigator's judgment for other reasons.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-08-23 (Actual); Primary Completion 2018-04-19 (Actual); Study Completion 2018-04-19 (Actual)

PRIMARY OUTCOMES:
Change from baseline in flow mediated dilatation | 4 weeks, up to maximum 5 weeks

SECONDARY OUTCOMES:
Rate of change from baseline in nytrotyrosine marker | 4 weeks, up to maximum 5 weeks
Rate of change from baseline in Intercellular Adhesion Molecule-1 | 4 weeks, up to maximum 5 weeks
Rate of change from baseline in Interleukin-6 | 4 weeks, up to maximum 5 weeks
Rate of change from baseline in C-reactive protein | 4 weeks, up to maximum 5 weeks
Change from baseline in blood pressure (irbesartan/atorvastatin fixed-dose combination group and irbesartan group) | 4 weeks, up to maximum 5 weeks
Change from baseline in low density lipoprotein-C (irbesartan/atorvastatin fixed-dose combination group and atorvastatin group) | 4 weeks, up to maximum 5 weeks
Change from baseline in total cholesterol (irbesartan/atorvastatin fixed-dose combination group and atorvastatin group) | 4 weeks, up to maximum 5 weeks
Change from baseline in high density lipoprotein-C (irbesartan/atorvastatin fixed-dose combination group and atorvastatin group) | 4 weeks, up to maximum 5 weeks
Change from baseline in triglycerides (irbesartan/atorvastatin fixed-dose combination group and atorvastatin group) | 4 weeks, up to maximum 5 weeks
Change from baseline in apolipoprotein-A1 (irbesartan/atorvastatin fixed-dose combination group and atorvastatin group) | 4 weeks, up to maximum 5 weeks
Change from baseline in apolipoprotein-B (irbesartan/atorvastatin fixed-dose combination group and atorvastatin group) - Time Frame: 4 weeks, up to maximum 5 weeks | 4 weeks, up to maximum 5 weeks
Percentage of participants with decreased level of blood pressure (irbesartan/atorvastatin fixed-dose combination group and irbesartan group) | 4 weeks, up to maximum 5 weeks
Rate of change from baseline in immunosenescence T cell fractionation | 4 weeks, up to maximum 5 weeks
Rate of change from baseline in T-cell induced inflammatory factors | 4 weeks, up to maximum 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org